CLINICAL TRIAL: NCT03539445
Title: Efficacy and Safety of Butylphthalide for Acute Ischemic Stroke Patients Receiving Intravenous Thrombolysis or Endovascular Treatment: A Prospective, Randomized, Double-blinded, Placebo Parallel Controlled, Multiple-center Trial.
Brief Title: Efficacy and Safety of Butylphthalide for Acute Ischemic Stroke Patients Receiving Intravenous Thrombolysis or Endovascular Treatment
Acronym: BAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Chief of Department of Neurological Intervention, Tian Tan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016YFC1301501
Record Dates: First submitted 2018-04-09; First posted 2018-05-29 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Acute Ischemic Stroke
Keywords: AIS; butylphthalide; mechanical thrombectomy; iv-rtPA; recovery of dysfunction
MeSH Terms: conditions — Ischemic Stroke | interventions — 3-n-butylphthalide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butylphthalide (Experimental): Drug: Butylphthalide Sodium Chloride Injection and Butylphthalide Soft Capsules
  Interventions: Drug: Butylphthalide
- Placebos (Placebo Comparator): Drug: Butylphthalide Placebo Injection and Butylphthalide Placebo Soft Capsules
  Interventions: Drug: Butylphthalide Placebo

INTERVENTIONS:
Drug: Butylphthalide — This group will receive a 3-month regimen of Butylphthalide and Sodium Chloride Injection 100ml twice/day in the initial 14 days and Butylphthalide Soft Capsules 0.2g triple/day for the rest Day 15 to Day 90.
  Other Names: dl-NBP
  Arms: Butylphthalide
Drug: Butylphthalide Placebo — This group will receive a 3-month regimen of Butylphthalide Placebo Injection 100ml twice/day in the initial 14 days and Butylphthalide Placebo Soft Capsules 0.2g triple/day for the rest Day 15 to Day 90.
  Other Names: Blank
  Arms: Placebos

SUMMARY:
Butylphthalide, as a well-known neuroprotective medication, is a family of compounds initially isolated from the seeds of Apium graveolens Linn, of which active ingredient is dl-3-N-butylphthalide (dl-NBP). With the significant effects of reducing the cerebral ischemic damage and eventually improving patients' clinical outcomes, by the potential mechanisms of promoting microcirculation, as well as releasing oxidative stress, mitochondrial dysfunction and poststroke inflammation, dl-NBP has been widely applied in acute ischemic stroke as an anti-ischemic drug in China since 2002. While with the evolution of using iv. recombinant tissue plasminogen activator（rtPA ）and mechanical thrombectomy in acute ischemic stroke（AIS）patients, it is still undefined whether combination therapy with dl-NBP could enhance the curative effect. The primary purpose of this trial is to evaluate the recovery of neurological deficits in AIS patients who receive iv-rtPA and/or mechanical thrombectomy with the a 3-month regimen of Butylphthalide and Sodium Chloride Injection 100ml twice/day in the initial 14 days and Butylphthalide Soft Capsules 0.2g triple/day for the rest 15th to 90th day therapy versus a 3-month regimen of Butylphthalide Placebo Injection 100ml twice/day in the initial 14 days and followed by Butylphthalide Placebo Soft Capsules 0.2g triple/day for the rest 15th to 90th day therapy.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, double-blinded, placebo parallel controlled, multiple-center trial. A total of approximately 1200 patients (Age≥18years) within 6 hours of symptom onset of acute ischemic stroke, who shows NIHSS from 4-25 points and intend to be treated with iv-rtPA and/or mechanical thrombectomy will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content, meanwhile the first injection will be within 6 hours from stroke onset : 1) one group will receive Butylphthalide and Sodium Chloride Injection 100ml twice/day in the initial 14 days, then take Butylphthalide Soft Capsules 0.2g triple/day for the rest 15th to 90th day therapy; 2) the other group will receive Butylphthalide Placebo Injection 100ml twice/day in the initial 14 days and then take Butylphthalide Placebo Soft Capsules 0.2g triple/day for the rest 15th to 90th day therapy. The primary objective is to explore whether the dl-NBP can improve the proportion of patients with a favorable outcome after receiving iv-rtPA and/or mechanical thrombectomy. The study consists of four visits including the day of randomization, 2 days after the first injection, 14 days when the injection therapy is done, and 30, 60 and 90 days when the oral therapy is finished. Demographic information, symptoms and signs, laboratory test, neuro-imaging assessment neurological function rating scale will be recorded during the program. The favorable outcome based on the 90-day modified Rankin Scale score was adjusted for baseline stroke severity, which was defined as a modified Rankin Scale score of 0 in patients with a baseline NIHSS core of 4 to 7, a modified Rankin Scale score of 0 to 1 in patients with a baseline NIHSS score of 8 to 14, and a modified Rankin Scale score of 0 to 2 in patients with a baseline NIHSS score of 15 to 25. The trial is anticipated to last from June 2018 to December 2022 with 1200 subjects recruited form 36 centers in China. All the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese Good Clinical Practice standard. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by Institutional Review Board (IRB) and Ethics Committee(EC) in Being Tiantan hospital, Capital Medical University.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged ≥ 18 years.
2. Acute ischemic stroke.
3. Within 6 hours from symptom onset.
4. Baseline NIHSS range 4 from 25.
5. Proceed to iv-rtPA or intravascular therapy including arterial thrombolysis and mechanical thrombectomy or bridging therapy.
6. Provision of informed consent.

Exclusion Criteria:

1. Modified Rankin Scale（mRS）>1 at randomization (pre-morbid historical assessment).
2. ASPECT ≤ 6 confirmed by the pre-operation CT scan.
3. Diagnosis of intracranial hemorrhagic disease, such as intracranial hemorrhage, subarachnoid hemorrhage and so on.
4. Use any drugs related to Butylphthalide during onset between randomization.
5. Dysphagia at the onset of stroke.
6. History of coagulation dysfunction, systemic bleeding, neutropenia or thrombocytopenia.
7. History of chronic hepatopathy, liver and kidney dysfunction, elevating Alanine transaminase (> 3 times normal upper limit), elevating serum creatinine (> 2 times normal upper limit).
8. History of severe cardio-pulmonary diseases which is not suitable for this study judged by investigator.
9. History of bradycardia (heart rate < 60 beats/m) and Sick sinus syndrome.
10. Severe non-cardiovascular comorbidity with life expectancy < 3 months or failed to follow the study for other reasons.
11. History of drug or food allergy, or are known to be allergic to the drug components of this study.
12. Contraindications for the digital subtraction angiography procedure, including severe allergy for contrast agent with or without Iodine.
13. Pregnancy or lactation, and women of childbearing age not practicing reliable contraception who do not have a documented negative pregnancy test.
14. Incapable to follow this study for mental illness, cognitive or emotional disorder.
15. Unsuitable for this study in the opinion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1216 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Favorable outcome | 90 days
  A modified Rankin Scale score of 0 in patients with a baseline NIHSS core of 4 to 7, a modified Rankin Scale score of 0 to 1 in patients with a baseline NIHSS score of 8 to 14, and a modified Rankin Scale score of 0 to 2 in patients with a baseline NIHSS score of 15 to 25.

SECONDARY OUTCOMES:
Neurological recovery | 90 days
  The difference value of the NIHSS between Day 14/Day 90 and the baseline
Cerebral infarction volume | 14 days
  Cerebral infarction volume at the Day 14 of the therapy
Recanalization rate | 24 hours
  Recanalization rate at the first 24 hours during the therapy
Symptomatic intracranial hemorrhage | 24 hours
  The percentage of symptomatic intracranial hemorrhage.
Recurrent stroke | 90 days
  New symptomatic vascular events (ischemic or hemorrhage) .
Recurrent ischemic stroke | 90 days
  Recurrent symptomatic ischemic stroke events
Any vascular complications | 90 days
  The quantity of patients who has complications with vascular events (recurrent symptomatic ischemic stroke, myocardiac infarction, vascular death)
EuroQol-5-Dimensions Scale（EQ-5D）questionnaire for measuring generic health status | 90 days
  Generic health status evaluated by EQ-5D questionnaire at the end of the therapy，which consists of two components：EuroQol-5-Dimensions Scale（EQ-5D）for health state description and Visual analogue scale（VAS）for self-evaluation. EQ-5D descriptive system covers five dimensions including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three response levels (no problem, some problems, and severe problems). The EQ-5D descriptive system generates 243 health states, each of which was assigned a utility score ranging from -0.59 to 1.00 (full health). While the EQ-5D also includes a 20-cm vertical VAS, with 0 and 100 representing worst and best imaginable health states, respectively. We classified the EQ-VAS scores into four groups, namely<65 (bad), 65 to 79 (fair), 80 to 89 (good), and 90 to 100 (excellent).
Cognitive function evaluated by the Mini-mental State Examination（MMSE） | 90 days
  Cognitive function evaluated by the Mini-mental State Examination（MMSE）at the end of the treatment，which effected by age and education experience. Cognitive impairment is diagnosed when MMSE ≤17 for illiteracy，MMSE ≤20 for those who take less than 6-years primary education，MMSE ≤24 for those have at least a middle school education.
Cognitive function evaluated by the Montreal Cognitive Assessment（MoCA） | 90 days
  Cognitive function evaluated by the Montreal Cognitive Assessment（MoCA） Scales at the end of the treatment, while taking MoCA <26 as cognitive impairment. Further more, when patient has a education experiment less than 12 years, investigator should give him or her one more score.
Favorable outcome | 14 days
  A modified Rankin Scale score of 0 in patients with a baseline NIHSS core of 4 to 7, a modified Rankin Scale score of 0 to 1 in patients with a baseline NIHSS score of 8 to 14, and a modified Rankin Scale score of 0 to 2 in patients with a baseline NIHSS score of 15 to 25.
Neurological recovery | 14 days
  The difference value of the NIHSS between Day 14/Day 90 and the baseline
Severity Adverse Event | 90 days
  The percentage of the Severity Adverse Events within the 14 days of the therapy.
Symptomatic intracranial hemorrhage | 90 days
  The percentage of symptomatic intracranial hemorrhage.
Total mortality | 90 days
  All deaths reported post-randomization will be recorded and adjudicated. Deaths will be subclassified by the adjudication committee as cardiovascular or non-cardiovascular.
Adverse Events | 90 days
  The percentage of the Adverse Events during the therapy.
Severity Adverse Event | 14 days
  The percentage of the Severity Adverse Events within the 14 days of the therapy.
Total mortality | 14 days
  All deaths reported post-randomization will be recorded and adjudicated. Deaths will be subclassified by the adjudication committee as cardiovascular or non-cardiovascular.
Adverse Events | 14 days
  The percentage of the Adverse Events during the therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang A, Jia B, Zhang X, Huo X, Chen J, Gui L, Cai Y, Guo Z, Han Y, Peng Z, Jing P, Chen Y, Liu Y, Yang Y, Wang F, Sun Z, Li T, Sun H, Yuan H, Shao H, Gao L, Zhang P, Wang F, Cao X, Shi W, Li C, Yang J, Zhang H, Wang F, Deng J, Liu Y, Deng W, Song C, Chen H, He L, Zhao H, Li X, Yang H, Zhou Z, Wang Y, Miao Z; BAST Investigators. Efficacy and Safety of Butylphthalide in Patients With Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2023 Aug 1;80(8):851-859. doi: 10.1001/jamaneurol.2023.1871. PMID 37358859
- [Derived] Zhang X, Wang A, Zhang JY, Jia B, Huo X, Zuo Y, Tian X, Wang Y, Miao Z; BAST study investigators. Efficacy and safety of butylphthalide for patients who had acute ischaemic stroke receiving intravenous thrombolysis or endovascular treatment (BAST trial): study protocol for a randomised placebo-controlled trial. BMJ Open. 2021 May 25;11(5):e045559. doi: 10.1136/bmjopen-2020-045559. PMID 34035100